CLINICAL TRIAL: NCT00813280
Title: Barriers to the Implementation of Complete Insulin Order Sets in the Management of Individuals With Hyperglycemia or Diabetes at Park Nicollet Methodist Hospital
Brief Title: Barriers to the Implementation of Complete Insulin Order Sets
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Park Nicollet Foundation (Other)
Responsible Party: Lisa Fish, MD
Other Study IDs: 03735-08-A
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2008-12

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hyperglycemia: hospitalized patients with BG >300 ml/dL

SUMMARY:
The major purpose of this Quality Improvement project is to begin to address the issues surrounding glycemic control in the hospital setting by collecting accurate, reliable and verifiable data on the occurrence of hyperglycemia (BG >300 mg/dL), and whether or not CIO is used (immediately before and 72 hours after the BG >300 mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* Park Nicollet Methodist Hospital patient
* recorded BG > 300 mg/dL during the study data collection period
* admitted to general floor hospital units

Exclusion Criteria:

* birth center
* intensive care units
* eating disorder unit
* pediatric patients < 18 years of age
* patients receiving insulin infusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with blood glucose >300 mg/dL
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
glucose levels | 72 hours

SECONDARY OUTCOMES:
type of insulin treatment | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fish, MD, Principal Investigator — Park Nicollet Health Services Endocrinology; Robert M Cuddihy, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- Park Nicollet Methodist Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Malmberg K, Ryden L, Efendic S, Herlitz J, Nicol P, Waldenstrom A, Wedel H, Welin L. Randomized trial of insulin-glucose infusion followed by subcutaneous insulin treatment in diabetic patients with acute myocardial infarction (DIGAMI study): effects on mortality at 1 year. J Am Coll Cardiol. 1995 Jul;26(1):57-65. doi: 10.1016/0735-1097(95)00126-k. PMID 7797776